CLINICAL TRIAL: NCT01241474
Title: Chronic Long-chain n-3 PUFA Supplement and Insulin Action in Human Subjects With Impaired Glucose Regulation
Brief Title: Effect of Fish Oil on Insulin Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UofAberdeen RINH HNU800
Record Dates: First submitted 2010-11-10; First posted 2010-11-16 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Metabolic Syndrome X; Type 2 Diabetes Mellitus; Sarcopenia
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus, Type 2; Sarcopenia | interventions — Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fish oil (Experimental)
  Interventions: Dietary Supplement: EPAX 6000 (marine omega 3 EPA/DHA fatty acid concentrates
- Maize (corn) oil (Placebo Comparator)
  Interventions: Dietary Supplement: Maize (corn) oil

INTERVENTIONS:
Dietary Supplement: EPAX 6000 (marine omega 3 EPA/DHA fatty acid concentrates — 6 x 1g capsules per day of marine oil (contains 3g/d docosahexaenoic acid plus eicosapentaenoic acid) for a 9 month period
  Other Names: EPAX 6000TG code F0-5222/XT
  Arms: Fish oil
Dietary Supplement: Maize (corn) oil — 6 x 1g capsules per day for 9 months
  Other Names: Banner chemicals product GL-518/XT
  Arms: Maize (corn) oil

SUMMARY:
The purpose of this study is to determine whether a prolonged (9 month) high (6g/d) of marine oil improves insulin sensitivity and glucose control in subjects with impaired glucose regulation.

DETAILED DESCRIPTION:
The incidence of Type 2 diabetes is related both to age and obesity. The disease impacts on quality of life and treatments represent a major health cost. Prevention or delayed onset of the disease remains a key target. Animal studies have shown that provision of high amounts of fish oil in the diet improves insulin sensitivity but human trials have proved equivocal. Recent dose-response trials in animals have shown the improved insulin sensitivity only occurs when the proportion of n-3 long chain polyunsaturated fatty acids (n-3 PUFA), docosahexaenoic acid and eicosapentaenoic acid, exceeds 14% of the total phospholipid fraction within tissue cell membranes. To achieve such values in humans would require a high dose of n-3 PUFA supplied over a prolonged period of time. This is tested within the current study where a daily dose of 6 g day of fish oil (containing a total of 3g docosahexaenoic acid plus eicosapentaenoic acid) is supplied for 9 months. As well as improving control of glycemia increased insulin sensitivity may also enhance protein metabolism and reduce the impact of frailty in older subjects.

ELIGIBILITY:
Inclusion Criteria:

* Men and post-menopausal women aged 40-65 years
* Recruited from the surrounding community of Aberdeen
* Insulin resistance with either

  1. venous plasma fasting glucose > 5.0, < 7.0 mmo/l,
  2. venous plasma 2-h 75-g OGTT > 5.0, < 11.1 mmol/l
  3. newly diagnosed with type 2 diabetes; must be asymptomatic and detected during our screenings and not require oral hypoglycemic or insulin therapy, HbA1c < 7.0%

Exclusion Criteria:

* Diabetes requiring oral hypoglycemic therapy or insulin
* Treatment with anticoagulants, regular steroids or non-steroidal anti-inflammatory drug treatment, tricyclic antidepressants, anti-arrhythmics
* Hepatic failure
* Renal failure
* Significant respiratory disease
* Anaemia
* Cardiovascular disease
* Malignancy
* Thromboembolic or coagulation disorders
* Alcoholism or other substance misuse
* Eating disorders or significant psychiatric disorders

Ages: 40 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change in insulin sensitivity assessed by hyperinsulinemic-euglycemic-eu-aminoacidemic clamp | 0 months and 9 months

SECONDARY OUTCOMES:
Change in amount of docosahexaenoic acid and eicosapentaenoic acid incorporated into phospholipid fraction of red blood cell membranes | at monthly intervals between 0 and 9 months
Change in plasma inflammatory markers | 0, 4 and 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Gerald E Lobley, BSc PhD, Principal Investigator — Rowett Institute of Nutrition and Health, University of Aberdeen
Locations (1):
- Rowett Institute of Nutrition and Health, University of Aberdeen, Aberdeen, United Kingdom